CLINICAL TRIAL: NCT05314725
Title: Treatment With SGLT-2 Inhibitor for Postoperative Hyperglycemia in Acute Abdominal Surgery - a Randomized Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-094-2021
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Hyperglycemia; Stress Hyperglycemia
Keywords: acute abdominal surgery; SGLT-2 inhibitor
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGLT-2 inhibitor (Experimental)
  Interventions: Drug: SGLT2 inhibitor
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGLT2 inhibitor — 10 days of SGLT2 inhibitor after surgery
  Arms: SGLT-2 inhibitor
Drug: Placebo — 10 days of placebo after surgery
  Arms: placebo

SUMMARY:
The aim of the study is to investigate the effect of an SGLT-2 inhibitor on postoperative hyperglycemia after acute abdominal surgery in patients without diabetes

ELIGIBILITY:
Inclusion Criteria:

* - Admitted to the ward after acute abdominal surgery (ASAP patient at Slagelse Hospital, OMEGA patient at Zealand University Hospital)
* At least two independent measurements of blood glucose above 7.7mmol/l within the first 48 hours after surgery
* Age of 18 to 85
* Must be able to understand and sign informed content

Exclusion Criteria:

* Patients diagnosed with diabetes mellitus

  * Impaired kidney function (eGFR < 45mL/min)
  * Severe liver disease (defined as transaminases above X 3 normal levels)
  * Acute pancreatitis within the last two months or a history of chronic pancreatitis
  * Participation in another pharmacological intervention trial
  * Predictable poor compliance (for instance mentally impaired)
  * Pregnancy or lactation (fertile women must have a negative serum or urine pregnancy test to participate)
  * Allergy to study medication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
time in range | from inclusion until 10 days after (or when the patient leaves the hospital)
  percentage of time in range defined as blood glucose between 3.9 and 7.8mmol/l. Blood glucose will be measures continuously while taking the study medication)

SECONDARY OUTCOMES:
mean glucose | from inclusion until 10 days after (or when the patient leaves the hospital)
glucose variability | from inclusion until 10 days after (or when the patient leaves the hospital)
  standard deviation divided by the mean and standard deviation
time with level 1 hypoglycemia | from inclusion until 10 days after (or when the patient leaves the hospital)
  blood glucose 3.0-3.9mmol/l
time with level 2 hypoglycemia | from inclusion until 10 days after (or when the patient leaves the hospital)
  blood glucose less than 3mmol/l
time with hyperglycemia | from inclusion until 10 days after (or when the patient leaves the hospital)
  blood glucose more than 10mmol/l
Quality of recovery-15 | every day while taking the study medication and on postoperative day 30
  Questionnaire assessing the patient's own sense of recovery after surgery
Nanostring | at inclusion, on day 4 of treatment and at end of treatment
  changes in up- and downregulation of genes

CONTACTS AND LOCATIONS:
Overall Officials: Emilie P Palmgren Colov, Principal Investigator — Zealand University Hospital

IPD SHARING:
Plan to Share IPD: No